CLINICAL TRIAL: NCT00276016
Title: Crossover Study of the Decongestant Effect of Phenylephrine Compared With Placebo and Pseudoephedrine as Active Control in SAR Subjects Exposed to Pollen in the Vienna Challenge Chamber
Brief Title: The Effects of Phenylephrine Compared With Those of Placebo and Pseudoephedrine on Nasal Congestion in Subjects With Seasonal Allergic Rhinitis (SAR)(P04579)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P04579
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Results first posted 2010-07-29 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Phenylephrine; Pseudoephedrine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Phenylephrine, Pseudoephedrine, Placebo (Experimental): Phenylephrine: Immediate-release 12 mg capsules for oral administration.
  Pseudoephedrine: 60 mg immediate-release tablets for oral administration.
  Placebo: Placebo capsules.
  Interventions: Drug: phenylephrine; Drug: pseudoephedrine; Drug: placebo
- Pseudoephedrine, Placebo, Phenylephrine (Experimental): Pseudoephedrine: 60 mg immediate-release tablets for oral administration.
  Placebo: Placebo capsules.
  Phenylephrine: Immediate-release 12 mg capsules for oral administration.
  Interventions: Drug: phenylephrine; Drug: pseudoephedrine; Drug: placebo
- Placebo, Phenylephrine, Pseudoephedrine (Experimental): Placebo: Placebo capsules.
  Phenylephrine: Immediate-release 12 mg capsules for oral administration.
  Pseudoephedrine: 60 mg immediate-release tablets for oral administration.
  Interventions: Drug: phenylephrine; Drug: pseudoephedrine; Drug: placebo
- Phenylephrine, Placebo, Pseudoephedrine (Experimental): Phenylephrine: Immediate-release 12 mg capsules for oral administration.
  Placebo: Placebo capsules.
  Pseudoephedrine: 60 mg immediate-release tablets for oral administration.
  Interventions: Drug: phenylephrine; Drug: pseudoephedrine; Drug: placebo
- Pseudoephedrine, Phenylephrine, Placebo (Experimental): Pseudoephedrine: 60 mg immediate-release tablets for oral administration.
  Phenylephrine: Immediate-release 12 mg capsules for oral administration.
  Placebo: Placebo capsules.
  Interventions: Drug: phenylephrine; Drug: pseudoephedrine; Drug: placebo
- Placebo, Pseudoephedrine, Phenylephrine (Experimental): Placebo: Placebo capsules.
  Pseudoephedrine: 60 mg immediate-release tablets for oral administration.
  Phenylephrine: Immediate-release 12 mg capsules for oral administration.
  Interventions: Drug: phenylephrine; Drug: pseudoephedrine; Drug: placebo

INTERVENTIONS:
Drug: phenylephrine — immediate-release 12 mg capsules for oral administration
Drug: pseudoephedrine — 60 mg immediate-release tablets for oral administration
Drug: placebo — placebo capsules

SUMMARY:
This is a Phase 3, single-dose, investigator-blind, randomized, placebo-controlled, crossover study, conducted at a single site in Austria, outside of the normal grass pollen season. An allergic reaction will be induced by exposing subjects to grass pollen in the Vienna Challenge Chamber (VCC). Subjects will receive a single dose of each of the following treatments according to a randomization sequence: Phenylephrine 12 mg immediate-release capsule, pseudoephedrine 60 mg immediate-release tablet, and placebo capsule. There will be a minimum of a 5-day washout period between each treatment. Subjects will complete symptom evaluations throughout the study. The nasal decongestant effects of phenylephrine will be compared to those of placebo using the subjective symptom evaluations. The safety profile (adverse events and vital signs) of the treatments will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Skin test positive for the grass pollen allergen used in the chamber at Screening or within the prior 12 months.
* A negative urine pregnancy test at Screening and at monthly intervals for female subjects of childbearing potential.
* The following minimum scores at an evaluation time point during each of the 120-minute screening period challenge sessions:

  1. Nasal Congestion Score of at least 2 (moderate);
  2. Total Nasal Symptoms Score of at least 6;
  3. Total Non-nasal Symptoms Score of at least 2.
* Freedom from any clinically significant disease, other than SAR, that would interfere with the study evaluations.

Exclusion Criteria :

* An upper or lower respiratory tract infection within 4 weeks before Screening.
* Dependence upon nasal, oral, or ocular decongestants, nasal topical antihistamines, or nasal steroids, in the opinion of the investigator.
* A known potential for hypersensitivity, allergy, or idiosyncratic reaction to the study drug or excipients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2006-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

REFERENCES:
- [Derived] Horak F, Zieglmayer P, Zieglmayer R, Lemell P, Yao R, Staudinger H, Danzig M. A placebo-controlled study of the nasal decongestant effect of phenylephrine and pseudoephedrine in the Vienna Challenge Chamber. Ann Allergy Asthma Immunol. 2009 Feb;102(2):116-20. doi: 10.1016/S1081-1206(10)60240-2. PMID 19230461

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject discontinued for reasons unrelated to treatment with study drug after the first dose (Intervention 1) of study drug Pseudoephedrine(PSE)
Period: Intervention 1
Arm/Group | Phenylephrine, Pseudoephedrine, Placebo | Pseudoephedrine, Placebo, Phenylephrine | Placebo, Phenylephrine, Pseudoephedrine | Phenylephrine, Placebo, Pseudoephedrine | Pseudoephedrine, Phenylephrine, Placebo | Placebo, Pseudoephedrine, Phenylephrine
Started | 7 | 7 | 7 | 6 | 6 | 6
Completed | 7 | 6 | 7 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Wash Out 1
Arm/Group | Phenylephrine, Pseudoephedrine, Placebo | Pseudoephedrine, Placebo, Phenylephrine | Placebo, Phenylephrine, Pseudoephedrine | Phenylephrine, Placebo, Pseudoephedrine | Pseudoephedrine, Phenylephrine, Placebo | Placebo, Pseudoephedrine, Phenylephrine
Started | 7 | 6 | 7 | 6 | 6 | 6
Completed | 7 | 6 | 7 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 2
Arm/Group | Phenylephrine, Pseudoephedrine, Placebo | Pseudoephedrine, Placebo, Phenylephrine | Placebo, Phenylephrine, Pseudoephedrine | Phenylephrine, Placebo, Pseudoephedrine | Pseudoephedrine, Phenylephrine, Placebo | Placebo, Pseudoephedrine, Phenylephrine
Started | 7 | 6 | 7 | 6 | 6 | 6
Completed | 7 | 6 | 7 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash Out 2
Arm/Group | Phenylephrine, Pseudoephedrine, Placebo | Pseudoephedrine, Placebo, Phenylephrine | Placebo, Phenylephrine, Pseudoephedrine | Phenylephrine, Placebo, Pseudoephedrine | Pseudoephedrine, Phenylephrine, Placebo | Placebo, Pseudoephedrine, Phenylephrine
Started | 7 | 6 | 7 | 6 | 6 | 6
Completed | 7 | 6 | 7 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 3
Arm/Group | Phenylephrine, Pseudoephedrine, Placebo | Pseudoephedrine, Placebo, Phenylephrine | Placebo, Phenylephrine, Pseudoephedrine | Phenylephrine, Placebo, Pseudoephedrine | Pseudoephedrine, Phenylephrine, Placebo | Placebo, Pseudoephedrine, Phenylephrine
Started | 7 | 6 | 7 | 6 | 6 | 6
Completed | 7 | 6 | 7 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenylephrine, Pseudoephedrine, Placebo | Pseudoephedrine, Placebo, Phenylephrine | Placebo, Phenylephrine, Pseudoephedrine | Phenylephrine, Placebo, Pseudoephedrine | Pseudoephedrine, Phenylephrine, Placebo | Placebo, Pseudoephedrine, Phenylephrine | Total
Number analyzed (Participants) | 7 | 7 | 7 | 6 | 6 | 6 | 39
Age, Customized [Mean (Standard Deviation); unit: years] | 27.9 (9.0) | 27.9 (3.3) | 24.9 (3.5) | 26.3 (1.6) | 28.0 (7.1) | 27.3 (3.3) | 27.0 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 1 | 3 | 5 | 23
  Male | 2 | 2 | 3 | 5 | 3 | 1 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Average Change From Baseline to Endpoint (6 Hours Post-dosing) in Nasal Congestion for Phenylephrine Compared With Placebo
Description: To evaluate the effect of phenylephrine 12-mg immediate-release capsule on nasal congestion in subjects with seasonal allergic rhinitis (SAR) who have been exposed to pollen for 6 hours in the Vienna Challenge Chamber (VCC). The average change from the Baseline was evaluated immediately before treatment start, over the first 6 hour post-dosing.
  The values for the scale are 0,1,2,3 for measure of symptoms, defined as 0-none, 1-mild, 2-moderate, 3-severe. They are subject-evaluated results.
Time Frame: Baseline to endpoint (6 hour period)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Phenylephrine
Number analyzed (Participants) | 38 | 38
Units on a scale
  Baseline score | 2.20 (0.36) | 2.20 (0.36)
  Change from Baseline to Endpoint Score | -0.12 (0.44) | -0.18 (0.44)
Statistical Analysis 1: Comparison: Placebo vs Phenylephrine; For endpoint; Test type: Superiority or Other; p = 0.561, ANOVA

2. Secondary Outcome: The Average Change From Baseline to Endpoint (6 Hours Post-dosing) in Nasal Congestion for Pseudoephedrine and Placebo.
Description: To estimate the effect of a pseudoephedrine (PSE) 60 mg immediate release tablet on nasal congestion over a 6-hour observation period relative to placebo
  The values for the nasal congestion score scale are 0,1,2,3 for measure of symptoms, defined as 0-none, 1-mild, 2-moderate, 3-severe. They are subject-evaluated results.
Time Frame: Baseline to endpoint (6 hour period)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pseudoephedrine | Placebo
Number analyzed (Participants) | 39 | 38
Units on a scale
  Baseline | 2.26 (0.36) | 2.20 (0.36)
  Endpoint | -0.47 (0.44) | -0.12 (0.44)
Statistical Analysis 1: Comparison: Pseudoephedrine vs Placebo; For endpoint; Test type: Superiority or Other; p < .001, ANOVA

ADVERSE EVENTS:
Arm/Group | Phenylephrine | Pseudoephedrine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less